CLINICAL TRIAL: NCT00497614
Title: 18F-FDG Positron Emission Tomography to Study the Response to Adalimumab in Rheumatoid Arthritis. A Monocentric Pilot Study
Brief Title: Positron Emission Tomography in Rheumatoid Arthritis With Adalimumab (PETRA)
Acronym: PETRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: University Hospital Tours
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOHP05-DM/PETRA
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2008-12-05 (Estimated); Status verified 2008-12

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Positron emission tomodensitometry; Tumor necrosis factor alpha inhibitor
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- No arm (Other)
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab

SUMMARY:
Biologics are routinely used for the treatment of rheumatoid arthritis (RA). Adalimumab is a human monoclonal antibody that inhibit the Tumor Necrosis Factor alpha (TNF-alpha). Identification of RA patients who respond to biologics is a challenging goal to avoid unnecessarily, costly and potentially harmful treatment.

The aim of the study is to address if 18 F FDG is a valuable biomarker for the assessment of the clinical response in RA with TNF-alpha blocking agent. Eight patients fulfilling the ACR (American College of Rheumatology) criteria will by enrolled. Patient will receive adalimumab according to the current guidelines i.e. 40mg /14 days sub cutaneously. The decision will stand on a high activity of the disease defined by the DAS 28 (Disease Activity Score) above 5.1. Positron emission tomography will be performed before, 2 and 12 weeks after the begin of the treatment. The response to adalimumab will by assessed by the SUV (standard Unit value) measured on the inflammatory joints of hands, wrist, ankle, feet and knees and compared to measurement of clinical (total swollen and tender joints count) echographic (synovium thickness and power doppler) and chemical biomarkers (erythrocyte sedimentation rate, C reactive protein).

ELIGIBILITY:
Inclusion Criteria: - Patients with active Rheumatoid arthritis PR définie selon les critères ACR (1987) (annexe 7) [18], Activité importante de la maladie (DAS 28 > 5,1) (annexe 5) [7], Indication d'un traitement par adalimumab (en accord avec l'A.M.M.), Homme ou femme dont l'âge est supérieur ou égal à 18 ans, Acceptant de participer à l'étude et ayant donné son consentement éclairé, Affiliés ou bénéficiaire d'un régime de sécurité sociale.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
There is no primary outcome measure specified for this study.

SECONDARY OUTCOMES:
There are no secondary outcome measures specified for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Denis Mulleman, MD, Principal Investigator — CHRU de Tours
Locations (1):
- University Hospital of Tours, Tours, France